CLINICAL TRIAL: NCT06948409
Title: The Choice of Neuromuscular Blockade Reversal Agent and Its Effects on Postoperative Urinary Retention: A Retrospective Cohort Study
Brief Title: NMBA Reversal and Postoperative Urinary Retention
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Luca J Wachtendorf, MD, Anesthesia Resident and Clinical Fellow, Co-Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 2025P000474; MISP #102761 (Other Grant/Funding Number: MERCK SHARP & DOHME LLC)
Record Dates: First submitted 2025-04-11; First posted 2025-04-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Neuromuscular Blocking Agents; Urinary Retention After Procedure; Urinary Retention Postoperative; Neuromuscular Blockade Reversal Agent; Neuromuscular Blockade; Costs; Atropine; Sugammadex; Glycopyrrolate; Neostigmine; Anesthesia
Keywords: Neuromuscular Blockade; Neuromuscular Blocking Agents; Sugammadex; Neuromuscular Blockade reversal agent; Urinary Retention Postoperative; Urinary Retention; Urinary Retention After Procedure; Costs; Neostigmine; Anesthesia; Atropine; Glycopyrrolate
MeSH Terms: conditions — Urinary Retention | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Choice of reversal agent (sugammadex or neostigmine [with muscaranic antagonist]) — The use of sugammadex or neostigmine (in co-administration with muscarinic antagonist) will be compared. The muscarinic antagonists that will be considered are atropine and glycopyrrolate.

SUMMARY:
In this single-center retrospective cohort study of adult patients who underwent surgery under general anesthesia at Beth Israel Deaconess Medical Center between September 2016 and January 2024, the association between the choice of neuromuscular blocking agent (NMBA) reversal strategy, comparing sugammadex with neostigmine (combined with a muscarinic antagonist), and postoperative urinary retention (POUR) will be evaluated. In secondary analyses, the effects of NMBA reversal strategy and POUR on costs of care and unplanned hospital visits will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Non-urinary system surgery
* General anesthesia
* Use of rocuronium or vecuronium for neuromuscular blockade
* Neuromuscular blockade reversal with sugammadex or neostigmine (with atropine and/or glycopyrrolate)
* Postoperative admission to the post-anesthesia care unit (PACU)

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≥ V
* Emergency reversal with sugammadex (≥ 16 mg/kg of sugammadex)
* Presence of foley or suprapubic catheter before or after the procedure
* Prior history of bladder resection surgery
* Observations with missing data for pre-specified confounding variables

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients at Beth Israel Deaconess Medical Center between September 2016 and January 2024
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2025-06-08 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
PACU discharge delay due to POUR | During the admission to the PACU (Perioperative, up to day 1)
  The primary outcome, post-anesthesia care unit (PACU) discharge delay due to postoperative urinary (POUR), will be defined as a documented delay in PACU discharge due to the inability to void. The PACU nurses or physicians responsible for immediate postoperative care routinely document these delays. Documentation about delays is required before a patient is discharged from the PACU. Within the individual categories "renal", "urinary", and "other", the investigators will search through all free text entries related to urinary retention. The study team will perform this review, and potential misspellings or synonyms will be identified and accounted for during the review process. The final primary endpoint, PACU discharge delay due to POUR, will be binary, and the endpoint data will be reported as frequency (total number [n] and proportion [%]).

SECONDARY OUTCOMES:
Costs of care | During the patient's hospital stay (Through study completion, an average of 1-2 weeks)
  Costs of care will be assessed using the hospital's cost calculations from an internal financial tracking system. This endpoint will include direct hospital costs, defined as variable and fixed costs directly associated with patient-care-related activities. To maintain the sensitive nature of cost data, the investigators will match the outcome data with data from the Healthcare Cost and Utilization Project-National Inpatient Sample (HCUP-NIS). Differences in total perioperative healthcare-associated costs in US-dollars between patients receiving different reversal strategies will be reported. While direct hospital cost data from the hospital network will serve as the outcome for linear regression analyses, the HCUP-NIS only provides total hospital costs. Thus, data will be matched with the HCUP-NIS data, and regression estimates from the study's dataset will subsequently be translated to obtain changes in total costs.
Unplanned hospital visits | Within 7 days after surgery
  Unplanned hospital visits within 7 days after ambulatory surgery will be defined as unplanned admission to the hospital after surgery, emergency department (ED) visits, or readmission to the hospital. Only patients undergoing ambulatory procedures will be included in this analysis. International Classification of Diseases, 10th Revision, Clinical Modification diagnostic codes, and notes related to the ED or readmission will be used to define unplanned hospital visits. Only the admission directly following the ambulatory procedure will be considered. If a patient undergoes more than one ambulatory procedure within 7 days before an inpatient admission, the procedure closest to the unplanned hospital visit will be identified as the index case.
Time to PACU discharge readiness | During the admission to the PACU (Perioperative, up to day 1)
  Time to PACU discharge readiness will be defined as the time from arrival to the PACU until a nurse has cleared the patient to be ready for discharge, measured in minutes. This outcome offers an accurate estimate of patient recovery independent from institutional factors such as bed availability or staffing, as opposed to the overall PACU length of stay.
PACU length of stay | During the admission to the PACU (Perioperative, up to day 1)
  PACU length of stay, measured in minutes, is the time between arrival until discharge from the PACU following surgery. In contrast to PACU discharge readiness, this endpoint considers the total time a patient spent in the PACU and correlates with the use of resources used (and subsequently costs) for post-anesthetic care for a patient.
Postoperative hospital length of stay | During the patient's hospital stay, defined as the time between surgery and day of discharge (Through study completion, an average of 1-2 weeks)
  Postoperative hospital length of stay will be defined as the time between surgery and discharge during the index hospitalization, measured in days. Patients undergoing ambulatory surgery will not be considered for this analysis.
Urinary catheter use or straight catheterization | Within 3 days after surgery
  The use of urinary catheters or straight catheterization within 3 days after surgery will be assessed. Patients undergoing ambulatory surgery will not be considered for this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian S Schaefer, MD, PhD, Principal Investigator — Center for Anesthesia Research Excellence, Beth Israel Deaconess Medical Center; Luca J Wachtendorf, MD, Principal Investigator — Center for Anesthesia Research Excellence, Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Due to the sensitive nature of the data collected for this study, requests to access the dataset from qualified researchers trained in human subject research and confidentiality may be sent to Maximilian S. Schaefer at msschaef@bidmc.harvard.edu.